CLINICAL TRIAL: NCT02329691
Title: Team, Competence and Safety Climate in the Operating Room
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Senior Consultant Surgeon, Associate professor, Sahlgrenska University Hospital
Other Study IDs: Team and safety
Record Dates: First submitted 2014-12-18; First posted 2015-01-01 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Surgery
Keywords: safety climate; surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Changes in the WHO checklist: Specific changes in the WHO checklist will be performed after observational studies to enhance the WHO checklist at the specific institution

SUMMARY:
The main objective is to explore and evaluate the effect of a change in the WHO checklist on the safety climate in the operating room at a University Hospital in Gothenburg.

DETAILED DESCRIPTION:
This study will assess the underlying safety climate in one operating ward at Sahlgrenska University Hospital, Göteborg. The Safety Attitude Questionnaire (SAQ) Operating Room version will be used to assess baseline safety climate. The use of the WHO check list will be investigated and documented according to a pre-defined CRF (case record form).

After this evaluation, changes in the WHO checklist will be performed. The changes will include educational efforts and involving focus groups to receive suggestions on improvements of the WHO checklist. The revised version of the WHO checklist will be implemented. To evaluate effects of the changes the SAQ will once again be distributed to the involved personnel.

The main objective is to explore, describe, educate and thereby improve the safety climate in the operating room. The setting is one of the operating room departments in Sahlgrenska University Hospital Gothenburg. The project includes to following parts:

* To assess baseline regarding the safety climate at a surgical ward at the Sahlgrenska University Hospital.
* Educational efforts on safety climate, team work, communication, and WHO check list by lectures and focus group discussions involving the OR team members to get input and suggestions on improvements of the WHO checklist.
* To explore differences in safety attitudes between different professions working in the OR.
* To identify areas for improvement in team work, communication and other non-technical skills.
* To re-implement the WHO check list with the aim to obtain more focus on the importance of teamwork and knowledge about the patient and procedure.
* To compare results from SAQ after implementation of safety related objectives with SAQ baseline data.

ELIGIBILITY:
Inclusion Criteria:

* Health care personnel working in the OR at Sahlgrenska University Hospital Östra, general surgery

Exclusion Criteria:

* All other health care personnel

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All health care personnel working in the OR at the general surgery department, Sahlgrenska University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Positive change in the Safety Attitudes Questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, Principal Investigator — Sahlgrenska Universitetssjukhuset/Östra
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

REFERENCES:
- [Derived] Erestam S, Haglind E, Bock D, Andersson AE, Angenete E. Changes in safety climate and teamwork in the operating room after implementation of a revised WHO checklist: a prospective interventional study. Patient Saf Surg. 2017 Jan 31;11:4. doi: 10.1186/s13037-017-0120-6. eCollection 2017. PMID 28163786